CLINICAL TRIAL: NCT03211728
Title: Does Perioperative Pregabalin Reduce Postoperative Pain After Arthroscopic Anterior Cruciate Ligament Reconstruction Surgery Under Spinal Anesthesia?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2017-0415
Record Dates: First submitted 2017-07-06; First posted 2017-07-07 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Anterior Cruciate Ligament (ACL) Reconstruction
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Intervention Model Description: Candidate for arthroscopic ACL reconstruction are divided into two groups of pregabalin and placebo with 48 patients in each group. The intervention group receive pregabalin 150 mg 1 hour before surgery and 12 hours after initial dose and a placebo is administered in control group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Drug: pregabalin
- placebo group (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pregabalin — The intervention group receive pregabalin 150 mg 1 hour before surgery and 12 hours after initial dose.
  Arms: experimental group
Drug: placebo — The placebo group receive placebo 150 mg 1 hour before surgery and 12 hours after initial dose.
  Arms: placebo group

SUMMARY:
The investigators hypothesize that perioperative oral administration of pregabalin would reduce postoperative pain and produce reduction in postoperative opioid consumption after anterior cruciate ligament (ACL) reconstruction . Patients are randomly assign to 1 of 2 groups. The placebo group receive placebo capsules 1 hour before surgery and 12 hours after initial dose. The pregabalin group receive pregabalin 150 mg, respectively at the same points.

ELIGIBILITY:
Inclusion Criteria:

* age between 20-65 years
* physical condition type I or II in ASA (American Society of Anesthesiology)

Exclusion Criteria:

* patients of ASA classification 3 or more
* with a history of cardiovascular or respiratory disease
* dizziness or frequent headache
* active alcohol or drug usage,
* intake of any analgesics daily or 48 hours before surgery
* impaired renal and/or hepatic function

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-08 (Actual)

PRIMARY OUTCOMES:
Postoperative pain scores | 12 hours after surgery
  Visual analog scale (VAS) score = 0-100 mm
Postoperative pain scores | 24 hours after surgery
  Visual analog scale (VAS) score = 0-100 mm
Postoperative pain scores | 36 hours after surgery
  Visual analog scale (VAS) score = 0-100 mm
Postoperative pain scores | 2 weeks after surgery
  Visual analog scale (VAS) score = 0-100 mm

SECONDARY OUTCOMES:
Opioid consumption | the first 48 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No